CLINICAL TRIAL: NCT02934152
Title: Symptom Assessment for Patients With Gastro-esophageal Reflux Disease Receiving Helicobacter Pylori Eradication
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201607055MINC
Record Dates: First submitted 2016-10-06; First posted 2016-10-14 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: Gastroesophageal reflux disease; Helicobacter pylori
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Rabeprazole; Amoxicillin; Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Early eradication (Experimental): Group A (H pylori eradication timing: early eradication, n=100): Initial H pylori eradication with triple therapy (rabeprazole 20 mg qd, amoxicillin 1gm bid, clarithromycin 500 mg bid) for two weeks.
  Interventions: Drug: H pylori eradication; Other: H pylori eradication timing
- Late eradication (Experimental): Group B (H pylori eradication timing: late eradication, n=100): PPI with rabeprazole 20 mg qd for 4 weeks, followed by H pylori eradication with triple therapy for two weeks
  Interventions: Drug: H pylori eradication; Other: H pylori eradication timing
- Negative Hp (Active Comparator): For patients with negative H. p infection documented by UBT (Group C, n=200), No H pylori eradication treatment will be given but PPI with rabeprazole 20 mg qd will be given for 8 weeks.
  Interventions: Drug: H pylori eradication

INTERVENTIONS:
Drug: H pylori eradication — H pylori eradication
  Other Names: rabeprazole, amoxicillin, clarithromycin
Other: H pylori eradication timing — Early or late eradication
  Arms: Early eradication; Late eradication

SUMMARY:
Background: Rebound acid hypersecretion and acid-related symptoms after discontinuation of proton-pump inhibitor has been reported in previous studies. In patients with concurrent gastro-esophageal reflux disease and Helicobacter pylori infection, whether eradication of H. pylori will aggravate acid-related symptoms after discontinuation of proton-pump inhibitor (PPI) remains elusive Objective: This study aims to investigate the incidence and severity of acid-related symptoms after discontinuation of proton-pump inhibitor in reflux patients receiving H. pylori eradication Expected result: The investigators will find out the incidence and severity of acid-related symptoms after discontinuation of proton-pump inhibitor in reflux patients receiving H. pylori eradication

DETAILED DESCRIPTION:
Background: Rebound acid hypersecretion and acid-related symptoms after discontinuation of proton-pump inhibitor has been reported in previous studies. In patients with concurrent gastro-esophageal reflux disease and Helicobacter pylori infection, whether eradication of H. pylori will aggravate acid-related symptoms after discontinuation of proton-pump inhibitor remains elusive Objective: This study aims to investigate the incidence and severity of acid-related symptoms after discontinuation of proton-pump inhibitor in reflux patients receiving H. pylori eradication Patients and methods: Consecutive reflux patients documented by validated questionnaires (GerdQ) and upper endoscopy will be enrolled from the outpatient clinic. After determination of H. pylori status by urea breath test (UBT), those with positive H. pylori infection will be randomized into two groups. Group A (n=100) will be given early H. pylori eradication with triple therapy for two weeks; group B (n=100) will be given rabeprazole 20 mg qd for 4 weeks, followed by H. pylori eradication with triple therapy for two weeks. The investigators will then determine the H. pylori status by urea breath test and the incidence and severity of acid-related symptoms with GerdQ at 4 weeks after H. pylori eradication. For patients with negative H. pylori infection (n=200), proton-pump inhibitor with rabeprazole 20 mg qd will be given for 8 weeks and the incidence and severity of acid-related symptoms will be evaluated with GerdQ at 4 weeks after discontinuation of PPI. The impact of H. pylori infection and H. pylori eradication and its timing on the incidence and severity of acid-related symptoms after discontinuation of proton-pump inhibitor will be analyzed.

Expected result: The investigators will find out the incidence and severity of acid-related symptoms after discontinuation of proton-pump inhibitor in reflux patients receiving H. pylori eradication

ELIGIBILITY:
Inclusion criteria:

1. Patients with typical reflux symptoms (heartburn and/or acid regurgitation) validated by standard questionnaire GerdQ.16
2. Aged >= 20 years old.
3. Willing to receive H. pylori eradication therapy.

Exclusion criteria:

1. Symptomatic reflux patients with high grade erosive esophagitis (LA classification Grade C and D) or Barrett's esophagus documented by endoscopy.
2. Symptomatic reflux patients with a history of using PPI in recent one month.
3. Subjects with known allergy to PPI.
4. Peptic ulcer disease
5. Cancers of the esophagus, stomach, and duodenum
6. Esophageal or gastric varices
7. Active upper gastrointestinal bleeding within 7 days prior to enrollment
8. Status after total or subtotal gastrectomy
9. Pregnancy
10. Use of anticoagulants or antiplatelets within one week prior to enrollment
11. Subjects with bleeding tendency

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2016-10; Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Acid rebound | 4 weeks
  Development of acid-related symptoms after discontinuation of proton-pump inhibitor in reflux patients receiving H. pylori eradication

SECONDARY OUTCOMES:
Severity of acid rebound | 4 weeks
  Severity of acid-related symptoms after discontinuation of proton-pump inhibitor in reflux patients receiving H. pylori eradication. The severity will be determined by the change of the scores of total and respective symptom items of the symptom questionnaire GerdQ.

CONTACTS AND LOCATIONS:
Overall Officials: Ping-Huei Tseng, MDPHD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hu KY, Tseng PH, Liou JM, Tu CH, Chen CC, Lee YC, Chiu HM, Wu MS. Rebound of Reflux-Related Symptoms After Helicobacter pylori Eradication in Patients With Gastroesophageal Reflux Disease: A Prospective Randomized Study. Helicobacter. 2025 Jan-Feb;30(1):e70023. doi: 10.1111/hel.70023. PMID 40007457